CLINICAL TRIAL: NCT05950555
Title: A Randomized, Double-blind Comparison of the Effects of Dexmedetomidine and Ketamine on Oxidative Stress Markers in Patients Under Combined Spinal-epidural Anesthesia Under Lower Extremity Surgery
Brief Title: The Effects of Two Anesthetic Drugs on Some Enzyme Levels in Patients Undergoing Lower Extremity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet AKSOY, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/23
Record Dates: First submitted 2023-06-05; First posted 2023-07-18 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Malondialdehyde; Heme Oxygenase; C-Reactive Protein
Keywords: Ketamine; Dexmedetomidine; Oxidative Stress; Antioxidant
MeSH Terms: interventions — Sodium Chloride; Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients given saline (Active Comparator): 10 cc/hour isotonic is given throughout the operation.
  Interventions: Other: Saline
- Patients given dexmedetomidine. (Active Comparator): Dexmedetomidine 0.1 µg/kg IV bolus followed by 0.2 µg/kg/hr infusion throughout surgery.
  Interventions: Other: Dexmedetomidine
- Patients given ketamine. (Active Comparator): Ketamine 0.2 mg/kg bolus followed by 0.1 mg/kg/hr infusion throughout surgery.
  Interventions: Other: Ketamine

INTERVENTIONS:
Other: Saline — We used 0.9% isotonic sodium chloride.
  Arms: Patients given saline
Other: Dexmedetomidine — We used the vial containing 200 mcg/2 ml i.v. concentrated infusion solution in 100 ml of 0.9% isotonic sodium chloride.
  Arms: Patients given dexmedetomidine.
Other: Ketamine — We used 500 mg/10 ml solution for injection in 0.9% isotonic sodium chloride.
  Arms: Patients given ketamine.

SUMMARY:
The primary aim of this study was to compare the effects of dexmedetomidine and ketamine, which are administered intravenously during surgery, on the levels of malondialdehyde, an antioxidant, anti-inflammatory enzyme, heme oxygenase-1 enzyme levels and C-reactive protein levels in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.

DETAILED DESCRIPTION:
This study was planned as double-blind; The researcher who evaluated the patient and recorded the data did not know which group the patient belonged to. The randomization sequence was generated with a computerized random number generator and patients were assigned to 3 groups, with 30 patients in each group.

The group to which the patient was included was listed in serially numbered sealed opaque envelopes. Another investigator (not involved in this study and not blinded to group assignment) administered CSEA to patients in a sitting position and opened the envelopes to see which group the patient belonged to, and prepared and administered the drugs to be used during anesthesia. An anesthetist, blinded to the group allocation, was responsible for collecting the intraoperative data. During and after surgery, data were recorded by and by this investigator. The blood of the patients was taken by the researcher who collected the data and delivered to the researchers who made the biochemical analyzes of their blood and blinded the groups. All surgeries were performed by the same surgical team and the same anesthesia team.

Peripheral IV vascular access was established using a 16/18-gauge cannula on the day of the operation. No premedication was applied to any patient before the operation. Before the anesthesia procedure, the patients' age, weight, height, body mass indexes, american society of anesthesiologists (ASA) physical status, systolic, diastolic and mean blood pressure baseline values, heart rate and oxygen saturation levels were recorded.

CSEA was applied to all patients in the sitting position. Following skin sterilization and local anesthetic infiltration (2% lidocaine), an 18-gauge Tuohy needle (CSEA, Braun, Melsungen, Germany) was advanced along the midline L3-4 or L4-5 intervertebral spaces using a loss of resistance technique. After negative pressure was detected, a 27-gauge pen-tipped spinal needle was inserted intrathecally using the needle-through-the-needle technique. After the free cerebrospinal fluid flow was observed, 1.8 ml 0.5% isobaric bupivacaine (9 mg) and 15 µg fentanyl were administered for 30 seconds. Then, the spinal needle was removed and the catheter was inserted into the epidural space, and it was advanced 3-5 cm in the space and controlled with negative pressure, and the catheter was fixed. At the end of the anesthesia procedure, the patients were placed in the supine position for the operation. The necessary study drugs were started to be administered to the patients in accordance with the study group they were assigned to, and infusions were continued throughout the operation.

The level of sensory block was assessed with the pinprick test, and surgery was allowed when the sensory block reached the upper level of the T12-L1 dermatome. If sensory block did not occur within the first 20 minutes following the spinal injection, spinal anesthesia was considered unsuccessful and the patients were excluded from the study. The patients who were excluded from the study were injected with an additional 5 ml of 2% lidocaine solutions through the epidural catheter until the sensory block T12-L1 level was achieved, and the patients were allowed to operate.

If the intrathecal space could not be reached in three unsuccessful attempts, a general anesthesia protocol was planned and patients requiring general anesthesia were excluded from the study.

For the measurement of MDA and HO-1 levels, blood samples taken from the patient groups included in the study were taken for 10-20 minutes for clotting. After the tube was kept in an upright position, it was centrifuged at +4°C at 4000 rpm for 15 minutes. The serum samples obtained were aliquoted and placed in a deep freezer at -80˚Ϲ and kept there until the day of analysis.

Serum malondialdehyde (MDA) and HO-1 levels were measured on the same day in order not to be affected by the variation between days. Serum MDA and HO-1 levels were determined by ELISA method, using "Human MDA ELISA Kit" and Human HO-1 ELISA Kit. measured in accordance with the manufacturer's instructions.

In addition, C-reactive protein (CRP) (mg/dl), calcium (mg/dl), alkaline phosphatase (U/L), lactate dehydrogenase (U/L), aspartate aminotransferase (U/L), alanine aminotransferase, which are routinely checked at preoperative, postoperative 2nd and 24th hours. (U/L), glucose (mg/dl), potassium (nmol/L), iron (ug/dl), total protein (g/dl) and albumin (g/dl) levels in Beckman Coulter device, ferritin (ng) /ml) Beckman Coulter device, Blood count parameters, White Blood Cell Count (10^3/mcL), Total Lymphocyte Count (10^3/mcL), Hemoglobin (g/dL) were studied on Sysmex device.

ELIGIBILITY:
Inclusion Criteria:

* ASA risk classification 1-2
* Patients who agreed to participate in the study

Exclusion Criteria:

* Body mass index (BMI) over 30 kg/m2
* Patients who will use bone cement in the surgical procedure
* Patients who will apply a tourniquet to the lower extremity
* Patients with vascular and coronary disease
* Patients with coagulation disorders that would prevent the application of CSEA
* Patients with allergies to the drugs to be used in the study
* Patients with increased head and intraocular pressure
* Patients with psychiatric and neuromuscular disorders
* Patients with multiple trauma
* Patients who did not consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Concentration of Malondialdehyde | just before surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on the level of malondialdehyde, which is an oxidative stress marker, in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.
Heme Oxygenase-1 | just before surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on the level of heme oxygenase-1, an antioxidant and anti-inflammatory enzyme, in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.
C-Reactive Protein | just before surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on C-Reactive Protein in patients undergoing lower extremity surgery under combined spinal epidural anesthesia.
Malondialdehyde | 2 hours after the start of surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on the level of malondialdehyde, which is an oxidative stress marker, in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.
Heme Oxygenase-1 | 2 hours after the start of surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on the level of heme oxygenase-1, an antioxidant and anti-inflammatory enzyme, in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.
C-Reactive Protein | 2 hours after the start of surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on C-Reactive Protein in patients undergoing lower extremity surgery under combined spinal epidural anesthesia.
Malondialdehyde | 24 hours after surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on the level of malondialdehyde, which is an oxidative stress marker, in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.
Heme Oxygenase-1 | 24 hours after surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on the level of heme oxygenase-1, an antioxidant and anti-inflammatory enzyme, in patients who underwent lower extremity surgery under combined spinal epidural anesthesia.
C-Reactive Protein | 24 hours after surgery
  The primary aim of this study was to investigate the effects of intravenous (iv) administration of dexmedetomidine and ketamine on C-Reactive Protein in patients undergoing lower extremity surgery under combined spinal epidural anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: İrfan Uç, Principal Investigator — Research Assistant
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we will decide later.